CLINICAL TRIAL: NCT02062983
Title: Early Predictor of Herceptin Cardio Toxicity in Breast Cancer Patients
Status: Suspended | Type: Observational
Why Stopped: Difficulty in enrolling patients
Sponsor: National Guard Health Affairs (Other Government)
Responsible Party: Sponsor
Other Study IDs: Herceptin
Record Dates: First submitted 2014-01-23; First posted 2014-02-14 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Herceptin: The study will be carried in prospective manner enrolling all patients diagnosed with breast cancer and over expressed human epidermal growth factor receptor 2 (HER2) and they are requiring Trastuzumab Neu adjuvant/ adjuvant /metastatic therapy as per standard care.
  Interventions: Drug: Herceptin

INTERVENTIONS:
Drug: Herceptin — Herceptin will be administered in different way per each setting as follow::total herceptin cycles are 18.
  Neu Adjuvant : chemo+herceptin, Surgery (hold herceptin) , Resume herceptin for 1 year period Adjuvant : Surgery, chemo+herceptin for 1 year period Metastatic : chemo+herceptin until progression.

SUMMARY:
Early identification of patients at risk for cardiotoxicity represent a primary goal for cardiologist and oncologist

From all adjuvant trials echocardiography is ideal for evaluating Left Ventricular function though its operator dependent. The use of other technique such as endomyocardial biopsy, is troublesome in clinical practice

Cardiac magnetic resonance imaging (MRI) have greater reproducibility in evaluating left ventricular ejection fraction (LVEF). This technique provides morphological, functional, perfusion, and viability information in one assessment. It is expensive and time consuming but id the diagnostic method of choice for patients with technically limited images from ECG and in patients with discordant information that is clinically significant from prior tests

DETAILED DESCRIPTION:
Current standard of care for patients while on adjuvant trastuzumab is baseline ECHO are as follows:

Patients on one of the above medications should undergo regular monitoring of the heart function during treatment as the following:

1. Baseline evaluation of LVEF prior inhibitor of therapy
2. Serial assessment of LVEF using the same modality.

There is no clear international guidelines on the frequency and method of LVEF assessment.

Cardiac function is usually measured by using (ECHO) echo cardiography and multiple-gated acquisition (MUGA) The patient should be assessed with the same techniques during treatment to avoid stressing the myocardium by the use of exercise or ionotropic agent, before measuring LVEF to prevent earlier evidence of cardiotoxicity. Changes in the early atrial (E/A) filling ratio reflect ventricular compliance and may predict diastolic dysfunction and so decline in LVEF.

Diastolic dysfunction seems to be predictive of cardiac morbidity and mortality.

Trials with adjuvant trastuzumab use the rules for stopping cardiotoxic agents. They identified subset of high risk patients by one or two of the following three criteria:

1. A decline with 10% or more in absolute LVEF from a normal base line to 50% or less
2. a high cumulative dose of Doxorubicin ( > 450 mg/m2 ) and / or;
3. abnormal baseline LVEF < 50% Patients who stopped taking doxorubicin after an LVEF decline were less likely to develop congestive heart failure (CHF) than those who did not.

Echocardiography is used regularly to monitor LVEF and is more widely available. The MUGA, in addition it does not expose patients to ionizing radiation but it is operator-dependent but training and use of automation may overcome the variation .

ELIGIBILITY:
Inclusion Criteria:

Breast cancer cases with histopathology prove of invasive carcinoma with HER 2 over expression detected by immunochemical stain and/ or FISH.

Age 18 to 80 years old. Patient with above criteria and eligible for Neu adjuvant/ adjuvant /metastatic( Trastuzumab) Herceptin therapy.

Normal blood count, liver function test and kidney function.

Exclusion Criteria:

Abnormal cardio vascular disease (ex. Heart Failure, Ischemic Heart Disease, post CABG) with EF≤50.

Valvular abnormality with reduced ejection fraction (EF). Recent Myocardiac Infraction / Ischemia Pregnancy or Breast feeding

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pilot study trying to identify early predictor for developing cardiotoxicity in such patients.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2012-06; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Estimate the incidence /of Herceptin induced heart failure in our population | 3 years
  To evaluate the reversibility of damage in patients on long term follow- up for a period of up to three years.
  To identify the applicability of troponin / cardiac natriuretic peptides (CNPS) as bio marker that can predict the occurrence of clinically significant left ventricular dysfunction.
  To evaluate the role of MRI in identifying patient at risk to develop cardio toxicity.
  Determine the frequency of elevated Troponin and B-type natriuretic peptide (BNP) in patient receiving adjuvant herceptin.

SECONDARY OUTCOMES:
Determine the incremental diagnostic value of Trop and BNP in predicting incidence of Hem CMP. | 3 years
  Determine the incremental diagnostic value of Trop and BNP in predicting incidence of Hem cardiac marker (CMP).
  Determine the relation between prior myocardial scaling and incidence of herceptin induced cardiac marker (CMP).
  Determine the correlation between myocardial edema, BNP and heart failure incidence of CMP

CONTACTS AND LOCATIONS:
Locations (1):
- National Guard Health Affairs, Riyadh, Riyadh Region, Saudi Arabia